CLINICAL TRIAL: NCT02531867
Title: A Multicenter, Post-Approval Clinical Study for Asfotase Alfa (Human Recombinant Tissue-nonspecific Alkaline Phosphatase Fusion Protein) Treatment for Patients With Hypophosphatasia (HPP) in Japan
Brief Title: Post-approval Clinical Study of Asfotase Alfa Treatment for Patients With Hypophosphatasia (HPP) in Japan
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AA-HPP-409
Record Dates: First submitted 2015-08-11; First posted 2015-08-25 (Estimated); Results first posted 2017-05-08 (Actual); Last update posted 2017-05-08 (Actual); Status verified 2017-03

CONDITIONS: Hypophosphatasia
Keywords: HPP; Bone Disease; Soft Bones; Low Alkaline Phosphatase; Genetic Metabolic Disorder; Alkaline Phosphatase; Rickets; Osteomalacia
MeSH Terms: conditions — Hypophosphatasia; Bone Diseases; Rickets; Osteomalacia | interventions — asfotase alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Asfotase Alfa (Experimental): Patients will receive asfotase alfa by subcutaneous injection. Asfotase alfa will be administered at either 2 mg/kg 3 times per week or 1 mg/kg 6 times per week depending on investigator's discretion.
  Interventions: Biological: Asfotase Alfa

INTERVENTIONS:
Biological: Asfotase Alfa
  Other Names: Strensiq

SUMMARY:
This is a multicenter study in Japan. Eleven sites which have already participated in the investigator-initiated clinical study (Early Access Program) will participate in this study.The objective of this study is to gain further information on the safety and efficacy of treatment with asfotase alfa.

DETAILED DESCRIPTION:
The primary objective of this study was to collect data on the safety of repeated subcutaneous (SC) injections of asfotase alfa. There were no secondary objectives. Exploratory objectives related to the efficacy of asfotase alfa are not being reported.

ELIGIBILITY:
Inclusion Criteria:

1. Patient or parent (or legal guardian) must provide written informed consent prior to the performance of any study-related procedures and must be willing to comply with study procedures. Where appropriate and required by local regulations, patient assent for participation must also be obtained.
2. Patient has completed the investigator-initiated clinical study (HPPJEAP-01) protocol for asfotase alfa

Exclusion Criteria:

1. Patient has a documented form of rickets caused by a condition other than HPP, including, but not limited to, rickets caused by 25(OH) vitamin D deficiency
2. Patient has serum calcium and/or phosphorus levels below the normal range
3. Patient is pregnant or lactating
4. Patient received treatment with bisphosphonates within 2 years prior to the Screening visit
5. Patient has a documented sensitivity to any of the components of asfotase alfa
6. Patient is currently enrolled in any other program or clinical study involving an investigational new drug, device, or treatment for HPP (eg, bone marrow transplantation)
7. Patient has clinically significant other disease in the opinion of the Investigator, defined as any other non HPP-related condition for which the patient is considered medically unstable.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenji Fujita, MD, Study Director — Medical Monitor

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 11 study sites, all in Japan; 13 patients were enrolled into this study. The first patient signed informed consent in June 2015; the study continued through November 2015 at multiple centers in Japan.
Groups:
- Overall Study: Patients enrolled in this study received a total of 6 mg/kg/week asfotase alfa by SC injection. At the Investigator's discretion, patients were continued on the dose established in the Investigator-initiated studies, receiving either 1 mg/kg asfotase alfa 6 times per week or 2 mg/kg asfotase alfa 3 times per week.
Period: Overall Study
Arm/Group | Overall Study
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All patients who met all of the inclusion and none of the exclusion criteria were considered the Baseline Analysis Population.
Arm/Group | Overall Study
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 1.39 [0.13 to 35.04]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 12
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) Including Injection Site Reactions (ISRs) and Injection Associated Reactions (IARs)
Description: Adverse events are any unwanted adverse medical occurrence in patients who are treated with a medicinal drug, whether or not considered drug-related. This includes events observed in patients administered with asfotase alfa between the first dose of asfotase alfa and the completion of patient's last visit for the clinical study.
Time Frame: Events that occurred between the first dose of asfotase alfa and the completion of the patient's last visit, which was up to 5 months.
Population: All patients who met all of the inclusion and none of the exclusion criteria were defined as the enrolled population, which was also the analysis population.The safety set comprised all patients who received at least 1 dose of the investigational drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 13
Participants
  Number of Patients with AEs | 9
  Number of Patients with ISRs | 2
  Number of Patients with IARs | 0

ADVERSE EVENTS:
Time Frame: Events that occurred between the first dose of asfotase alfa and the completion of the patient's last visit, which was up to 5 months.
Description: TEAEs were collected at every visit and follow-up.
Arm/Group | Overall Study
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 9/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Study (N=13)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Injection site bruising (General disorders) | 1 (1)
Injection site erythema (General disorders) | 1 (3)
Injection site induration (General disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Conjunctivitis viral (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (3)
Upper respiratory tract infection (Infections and infestations) | 2 (5)
Viral rash (Infections and infestations) | 1 (1)
Feeding tube complicatino (Injury, poisoning and procedural complications) | 1 (1)
Intercostal neuralgia (Nervous system disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigators are subject to certain disclosure and publication limitations. In cases of publication of the study results at conferences or on academic journals, the post-approval clinical study coordinating investigator and the study sponsor should discuss about details of publication, publication methods and presenters before decision-making